CLINICAL TRIAL: NCT05302245
Title: Caring Forward: A Longitudinal Examination of Unpaid Caregivers of Acquired Brain Injury (ABI) Survivors in Nova Scotia
Brief Title: A Longitudinal Examination of Unpaid Caregivers of Acquired Brain Injury (ABI) Survivors in Nova Scotia
Acronym: CaringForwrd
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Other Study IDs: 1025568; 1025253 (Other: IWK Health Centre REB Approval #)
Record Dates: First submitted 2021-03-15; First posted 2022-03-31 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Caregivers
Keywords: Caregivers; Acquired brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Caregivers of ABI survivors: Unpaid caregivers of acquired brain injury survivors living in Nova Scotia

SUMMARY:
The purpose of the present study is to follow unpaid caregivers of ABI survivors in Nova Scotia over time to learn more about their experiences. The study is funded by the Government of Nova Scotia (i.e. Department of Health and Wellness). The present longitudinal cohort study will help increase knowledge about ABI caregivers at a provincial level. Findings will also be used in developing future interventions to help caregivers in this population.

The goals of the research study are:

1. To understand the natural experiences of unpaid caregivers over time. More specifically, the investigators hope to learn about the experiences of unpaid caregivers of acquired brain injury survivors in Nova Scotia.
2. To examine the connection between study demographic variables (e.g. the amount of time spent caregiving in hours per week), and psychological outcome variables (e.g. caregiver burden).
3. To learn about the relationship between psychological outcome variables (e.g. psychological distress and savouring).
4. To provide a platform for future studies using the Trials within Cohort (TwiC) study design.

DETAILED DESCRIPTION:
The Investigators are employing a Trials within Cohorts research design. That is, they are conducting a prospective longitudinal cohort study, with the cohort serving as a platform in which future studies or interventions can be tested. In accordance with this approach, eligible participants who have given consent to be contacted in the future may be selected and approached for future participation in randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an unpaid, informal, caregiver of an ABI survivor
* Participant live in Nova Scotia
* Participant is able to read, write and understand English
* Participant has access to a tablet, smart phone, or computer with high speed internet
* Participant consents to complete online study questionnaires

Exclusion Criteria:

* Participant is a paid, professional caregiver of an ABI survivor
* Participant does not live in Nova Scotia
* Participant is not able to read, write and understand English
* Participant does not have access to a tablet, smart phone, or computer with high speed internet
* Participant does not consent to complete online study questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caregivers of ABI survivors living in Nova Scotia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Psychological strain | At baseline.
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | Six months following baseline.
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | Twelve months following baseline.
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | Eighteen months following baseline.
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).
Psychological strain | Twenty four months following baseline.
  The Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), a 21-item self-report measure that will assess caregiver's levels of psychological strain over the last week in three distinct categories; depression (e.g. hopelessness, depressed mood), anxiety (e.g. fear, anticipation of negative events), and stress (e.g. prolonged state of arousal, difficulty relaxing).

SECONDARY OUTCOMES:
Caregiver's perception of brain injury services in the community | At baseline.
  Services Obstacles Scale (SOS; Kolakowsky-Hayner et al., 2000), a 6-item scale that will be used to assess caregivers' perceptions of brain injury services in the community. The scale has three main components upon which the questions are based: 1) satisfaction with treatment resources; 2) finances as an obstacle to receiving services; and 3) transportation as an obstacle to receiving services.
Caregiver's perception of brain injury services in the community | Six months following baseline.
  Services Obstacles Scale (SOS; Kolakowsky-Hayner et al., 2000), a 6-item scale that will be used to assess caregivers' perceptions of brain injury services in the community. The scale has three main components upon which the questions are based: 1) satisfaction with treatment resources; 2) finances as an obstacle to receiving services; and 3) transportation as an obstacle to receiving services.
Caregiver's perception of brain injury services in the community | Twelve months following baseline.
  Services Obstacles Scale (SOS; Kolakowsky-Hayner et al., 2000), a 6-item scale that will be used to assess caregivers' perceptions of brain injury services in the community. The scale has three main components upon which the questions are based: 1) satisfaction with treatment resources; 2) finances as an obstacle to receiving services; and 3) transportation as an obstacle to receiving services.
Caregiver's perception of brain injury services in the community | Eighteen months following baseline.
  Services Obstacles Scale (SOS; Kolakowsky-Hayner et al., 2000), a 6-item scale that will be used to assess caregivers' perceptions of brain injury services in the community. The scale has three main components upon which the questions are based: 1) satisfaction with treatment resources; 2) finances as an obstacle to receiving services; and 3) transportation as an obstacle to receiving services.
Caregiver's perception of brain injury services in the community | Twenty four months following baseline.
  Services Obstacles Scale (SOS; Kolakowsky-Hayner et al., 2000), a 6-item scale that will be used to assess caregivers' perceptions of brain injury services in the community. The scale has three main components upon which the questions are based: 1) satisfaction with treatment resources; 2) finances as an obstacle to receiving services; and 3) transportation as an obstacle to receiving services.
Social support | At baseline.
  The Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988), a 12-item scale that will assess caregivers' perceived social support from three sources; family, friends, and a significant other.
Social support | Six months following baseline.
  The Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988), a 12-item scale that will assess caregivers' perceived social support from three sources; family, friends, and a significant other.
Social support | Twelve months following baseline.
  The Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988), a 12-item scale that will assess caregivers' perceived social support from three sources; family, friends, and a significant other.
Social support | Eighteen months following baseline.
  The Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988), a 12-item scale that will assess caregivers' perceived social support from three sources; family, friends, and a significant other.
Social support | Twenty four months following baseline.
  The Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988), a 12-item scale that will assess caregivers' perceived social support from three sources; family, friends, and a significant other.
Savouring | At baseline.
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | Six months following baseline.
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | Twelve months following baseline.
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | Eighteen months following baseline.
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Savouring | Twenty four months following baseline.
  The Savouring Configuration Inventory (SCI; Lauzon & Green-Demers, 2020), which measures hedonic savouring, and eudaimonic savouring of meaning of life, spirituality, self-reflection, inspiration, appreciation, and gratitude. It comprises 28 scenarios (4 subscales), paired with a single item.
Overall quality of life and general health | At baseline.
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | Six months following baseline.
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | Twelve months following baseline.
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | Eighteen months following baseline.
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Overall quality of life and general health | Twenty four months following baseline.
  The World Health Organization Quality of Life Assessment -BREF (WHOQOL-BREF; Whoqol Group, 1998), a 26-item measure that assesses quality of life in four distinct domains: physical health, psychological health, social relationships and the environment. A weighted summary score from 0-100 is calculated for each domain, with higher scores indicating higher quality of life.
Caregiver burden | At baseline.
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | Six months following baseline.
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | Twelve months following baseline.
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | Eighteen months following baseline.
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiver burden | Twenty four months following baseline.
  The Zarit Burden Interview-Short Form (ZBI-SF; Bedard et al., 2001), a 12-item measure that assesses individuals' perceived burden of providing care to their loved one.
Caregiving self-efficacy | At baseline.
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | Six months following baseline.
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | Twelve months following baseline.
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | Eighteen months following baseline.
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.
Caregiving self-efficacy | Twenty four months following baseline.
  The Controlling Upsetting Thoughts about Caregiving subscale from the 15-item Revised Scale for Caregiving Self-Efficacy (RSCSE; Steffen et al. 2002), that measure caregivers level of confidence with higher scores indicating higher levels of self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to indicate during Informed Consent whether their de-identified data may be shared with other researchers, provided the study is approved by an ethics board and researchers agree to use the data only for the purposes described in the approved research study. De-identified data from all outcome measures will be made available to approved researchers upon request, provided individual participants have provided consent.
Supporting Information: Study Protocol, SAP, ICF